CLINICAL TRIAL: NCT06154239
Title: Screening With Tampons: Evaluating Diagnostic Accuracy for STIs, BV and HPV and Assessing Participant Views
Brief Title: Screening With Tampons: Evaluating Diagnostic Accuracy and HPV and Assessing Participant Views
Acronym: STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne's Day Ltd (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LH-DA-01
Record Dates: First submitted 2023-11-08; First posted 2023-12-04 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chlamydia; Gonorrhea; Bacterial Vaginosis; Human Papilloma Virus
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Vaginosis, Bacterial

STUDY DESIGN:
Intervention Model Description: MAIN STUDY:
  All participants will have 3 samples taken: DAYE Diagnostic Tampon (DDT), self-swab and clinician administered swab. Participants will be randomised into 2 groups for sampling order between the DDT and self-swab.
  SUB-STUDY
  In the sub-study will only perform the DDT and self-swab. Participants will be randomised according to sample order for the DDT and self-swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A: Self-swab then DDT (Other): Participants will take the self-swab sample, followed by the DDT sample at home. They will then have the clinician swab taken in the clinic.
  Interventions: Device: DAYE Diagnostic Tampon; Diagnostic Test: Vaginal self-swab; Diagnostic Test: Clinician vaginal swab
- Arm B: DDT then self-swab (Other): Participants will take the DDT sample, followed by the self-swab sample at home. They will then have the clinician swab taken in the clinic.
  Interventions: Device: DAYE Diagnostic Tampon; Diagnostic Test: Vaginal self-swab; Diagnostic Test: Clinician vaginal swab
- Sub-study: Arm A: Self-swab then DDT (Other): Participants will take the self-swab sample, followed by the DDT sample at home.
  Interventions: Device: DAYE Diagnostic Tampon; Diagnostic Test: Vaginal self-swab
- Sub-study: Arm B: DDT then self-swab (Other): Participants will take the DDT sample, followed by the self-swab sample at home.
  Interventions: Device: DAYE Diagnostic Tampon; Diagnostic Test: Vaginal self-swab

INTERVENTIONS:
Device: DAYE Diagnostic Tampon — The DAYE Diagnostic Tampon is a class A in vitro diagnostic device. It has CE certification (self-certified via a declaration of conformity, following the IVDR (EU) 2017/746). The DDT is constructed entirely from woven cotton and consists of an absorbent core wrapped in a protective sleeve. The DDT is loaded in an applicator to aid with insertion.
Diagnostic Test: Vaginal self-swab — A vaginal self-swab typically consists of a long, slender, and flexible stick or handle, often made of plastic or a similar material. At one end, there's a soft, absorbent tip made of cotton or synthetic material. This tip is designed to collect a sample from the vaginal walls or cervix.
Diagnostic Test: Clinician vaginal swab — A clinician vaginal swab is a medical tool used by healthcare professionals to collect samples from the vaginal canal for diagnostic purposes. It's typically a long, thin, and flexible instrument. At one end, there's a cotton, rayon, or synthetic tip designed to collect cells, discharge, or other materials from the vaginal walls, cervix, or other areas within the vaginal canal.
  The clinician swab is not taken in sub-study participants.
  Arms: Arm A: Self-swab then DDT; Arm B: DDT then self-swab

SUMMARY:
Diagnostic trial comparing the diagnostic accuracy of the DAYE Diagnostic Tampon (DDT) with a vaginal swab (self-collected and clinician taken).

DETAILED DESCRIPTION:
MAIN STUDY DESIGN

A diagnostic trial comparing the diagnostic accuracy, usability and acceptability of the DAYE Diagnostic Tampon (DDT) compared to standard vaginal self-swabs and clinician administration of a vaginal swabs. Diagnostic accuracy will be compared for detection of Chlamydia, Gonorrhoea, BV & HPV.

A total of 350 eligible participants will be enrolled into the trial in the UK and Italy. To adequately assess DDT performance on specificity and sensitivity, participants will be recruited from one of two groups:

* Group 1: 50 participants with a recent confirmed HPV diagnosis (UK and Italy)
* Group 2: 300 participants from the general population (UK only)

All participants will be randomised according to sample order for the DDT and self-swab using block randomisation:

* Group A: Approximately half the participants will perform the self-swab followed by the DDT.
* Group B: Approximately half the participants will perform the DDT followed by the self-swab

All eligible participants will be provided with a trial kit containing the DDT and self-swab and attend at least 1 clinic visit as part of their participation in the trial. Participants will also provide answers to questionnaires at baseline and after all sampling is complete.

Participation in the trial is expected to last approximately 2-3 weeks (dependent on timing of clinic appointment(s)). All samples collected during the trial will be sent to a central laboratory for analysis, either in the UK or Italy i.e., samples will be analysed in the country they were collected.

SUB-STUDY DESIGN

A maximum of 210 eligible participants will be recruited and provide 2 samples to a decentralised sub-study to assess the DDTs performance compared to a self-taken vaginal swab. Recruitment will be stopped as soon as 21 positive cases of STI are confirmed by the lab.

* Group 3: 210 participants with suspected or recently confirmed chlamydia or gonorrhoea.

All participants will be randomised according to sample order for the DDT and self-swab using block randomisation:

* Group A: Approximately half the participants will perform the self-swab followed by the DDT.
* Group B: Approximately half the participants will perform the DDT followed by the self- swab

Pre-screening, informed consent, screening and eligibility assessments will occur online. Trial team will confirm e-consent and eligibility. Randomisation will be performed at the point of enrolment by a member of the trial team using a re-generated list of treatment allocation blocks. Some demographic information and medical history will be collected at baseline. All eligible participants will be provided with a trial kit containing the DDT and self-swab which they will use at home and send directly to the testing laboratory. Participants will also provide answers to questionnaires at baseline and after all sampling is complete. Participants will enter data directly into the EDC platform. Participation in the sub-study is expected to last approximately 1 week. All samples collected during the trial will be sent to a central accredited laboratory(s) for analysis in the UK.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 25-65 years.
2. People assigned female at birth (AFAB).
3. Sexually active individuals. In this case, "sexually active" is defined as having penetrative vaginal sex.
4. Group 1 only: Confirmed HPV+ diagnosis within the past 4 weeks.

   a. UK only: Ability to upload evidence of this diagnosis to the trial ePRO system (e.g. via a screenshot of the NHS app, or similar to be reviewed by the trial team).
5. Willingness to give informed consent and adhere to trial procedures.

Exclusion Criteria:

1. Previous hysterectomy or total hysterectomy with removal of cervix
2. Known allergy or sensitivity to tampons
3. History of TSS (both tampon-associated and non-tampon associated)
4. Individuals who are pregnant or breastfeeding.
5. Participation in another interventional clinical trial or use of investigational drugs in the last 30 days.
6. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial. -

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Evaluate the diagnostic accuracy of the Daye Diagnostic Tampon for detecting Chlamydia, Gonorrhea, BV and HPV | Within 4 weeks of the samples being received at the lab.
  Accuracy of the STI, BV and HPV detection using menstrual tampons compared to other specimen collection methods (clinician taken and self-swab) via assays

SECONDARY OUTCOMES:
Assess the usability of the DDT (via After-Scenario Questionnaire - ASQ) | Post-sampling (once all samples are collected) - at study completion usually after 4 weeks
  After scenario questionnaire scores - higher scores = more usable
Explore participants views of the usability and acceptability of the DDT | Pre-sampling (baseline) and Post-sampling (once all samples are collected) - at study completion usually after 4 weeks
  Quantitative and qualitative feedback from pre- and post-sampling questionnaires
Explore participants views of the usability and acceptability of the DDT | Through study completion, an average of 4-6 weeks
  Qualitative feedback from focus groups
Assess whether the DDT is a preferred sampling method for participants | Pre-sampling (baseline) and Post-sampling (once all samples are collected) - at study completion usually after 4 weeks
  User preferences (self-report)
Assess if the order of sample collection (self-swab vs DDT) impacts diagnostic accuracy as assessed by assays | Post sample analysis - 4 weeks after the last samples are received at the lab
  Comparison between the detection accuracy of infections between sample order (Group A and Group B) using assays
willingness to pay | Post-sampling (once all samples are collected) - at study completion usually after 4 weeks
  Willingness to pay for the DDT via questions in post-sampling questionnaire
Understand the health economic consequences of using the DDT for STI, BV and HPV testing - time taken | Post-sampling (once all samples are collected) - at study completion usually after 4 weeks
  Comparison of time taken for DDT vs clinician swab
Explore stakeholder attitudes to tampons as a means of sample collection for microbial testing. | Throughout the trial (and once stakeholders with a role in the trial have engaged with the tampon)
  Qualitative feedback from stakeholder questionnaires
Assess the occurrence of AEs/SAEs as a result of tampon sampling. | None expected, but any events will be collected and recorded on an ongoing basis as outlined in the protocol and analysed at study completion usually after 4 weeks
  AE/SAE occurrence.

OTHER OUTCOMES:
Explore the relationship between duration of wear and diagnostic accuracy. | Post sample analysis - 4 weeks after the last samples are received at the lab
  Duration of DDT wear and diagnostic accuracy
Sub-study Objective: Evaluate the diagnostic accuracy of the Daye Diagnostic Tampon for detecting STIs (Chlamydia, Gonorrhoea) specifically demonstrating a sensitivity of more than 70% for DDT. | Samples will be analysed around 2 weeks after collection. The outcome will be assessed as soon as 21 positive samples have been obtained.
  Accuracy of the STI detection using menstrual tampons compared to other specimen collection methods (self-swab) via Hologic APTIMA AC assay

CONTACTS AND LOCATIONS:
Overall Officials: Luke Twelves, Principal Investigator — Lindus Health
Locations (1):
- Lindus Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No